CLINICAL TRIAL: NCT00042367
Title: Pilot Study of Systemic and Intrathecal Chemotherapy Followed by Conformal Radiation for Infants With Brain Tumors
Brief Title: Study of Systemic and Spinal Chemotherapy Followed by Radiation for Infants With Brain Tumors
Acronym: BB'98
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Duke University (Other); St. Jude Children's Research Hospital (Other); Children's National Research Institute (Other); Seattle Children's Hospital (Other); Children's Hospital of Philadelphia (Other); University of Pittsburgh (Other); Dana-Farber Cancer Institute (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Susan Blaney, Professor of Pediatrics, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H8619; NCT00005063 (obsolete NCT alias)
Record Dates: First submitted 2002-07-26; First posted 2002-08-01 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Brain Tumors
MeSH Terms: conditions — Brain Neoplasms | interventions — Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Induction therapy (Regimen 1, Course 1, Cycle A1 — 2-8 hrs: Cisplatin 3.5 mg/kg + mannitol 0.4 g/kg in D5 NS (1000 ml/m2) over 6 hrs at approximately 167ml/m2/hr. 8-12 hrs: D5 NS (665 ml/m2) + KCl (2 mEq/100 ml) +MgSO4 (0.5 mEq/100 ml) at approximately 167ml/m2/hr.
  12-24 hrs: D5 NS + KCl (2 mEq/100 ml) + MgSO4 (0.5mEq/100 ml) at approximately 65 ml/m2/hr.
  Days 2,3: 0 hrs: Mesna 6 mg/kg IV in 0.65 ml/kg of IVF over 15 min 15 min: Cyclophosphamide 30 mg/kg IV over 30 min 45 min: Post-chemotherapy hydration - D5 1/2 NS + KCl(1 mEq/100 ml) at approximately 130 ml/m2/hr for at least 24 hours.
  3 hrs: Mesna 6 mg/kg IV in 0.65 ml/kg IVF over 15 min 6 hrs: Mesna 6 mg/kg IV in 0.65 ml/kg IVF over 15 min 9 hrs: Mesna 6 mg/kg IV in 0.65 ml/kg IVF over 15 min 12 hrs: Mesna 6 mg/kg IV in 0.65 ml/kg IVF over 15 min Day 4 G-CSF 5 µg/kg subcutaneously, daily until ANC ≥ 2000 on two consecutive days, post ANC nadir.
  Day 8: Vincristine 0.05 mg/kg IV push (max dose = 2 mg) Day 15: Vincristine 0.05 mg/kg IV push (max dose = 2 mg)
Drug: Regimen 1, Course 1, Cycle A2 (Days 22 - 42) — Drugs and doses are same as in Cycle A1. Cycle A2 begins following recovery from Cycle A1, but no sooner than day 21. Patients with delays in recovery beyond day 28 should have dose modifications
Drug: Cycle B — Days 43 - 63) Etoposide, 1.7 mg/kg p.o. qd x 21 days. The dose will be diluted immediately prior to administration in juice flavored syrup to a final concentration of 0.4 Each dose should be aken 1 hour before or 2 hours after a meal.
  Cycle B begins following recovery from Cycle A2; however, it begin no sooner than 21 days after the start of Cycle A2.
  Monitor weekly CBC/diff/plt. If ANC < 500/mm3 or platelets (unsupported) < 50,000/mm3 then discontinue etoposide. A 25% reduction should be made for the next cycle of oral etoposide.
  Interim Response Evaluation (Days 64 - 70) Interim Response Evaluation should be performed the week following the completion of Course 1.
Drug: Regimen 1, Course 2 — 6.3.3 Regimen 1, Course 2 Repeat systemic therapy as per Course 1 (Cycle A1, Cycle A2, and Cycle B) in patients with SD or better at the interim response evaluation (see Figure 2 for IT mafosfamide guidelines). Course 2 should not begin any sooner than 7 days after the completion of Course 1.
Drug: Intrathecal Mafosfamide — Regimen 1, Course 1 Mafosfamide, 14 mg, is given two times/week during Cycle A1 and Cycle A2 of Course 1, for 12 total doses during days 1-41. The first dose of Cycles A1 and A2 should be given, if possible, on the same day as the first I.V. cyclophosphamide dose and the second dose 3 to 4 days later. The assigned dose is given one time/week during Cycle B, Course 1 for 3 total doses during days 43 - 63.
Drug: Regimen 1 Course 2, IT mafosfamide — Regimen 1, Course 2 The assigned dose is administered once with IV cyclophosphamide during each of Cycle A1 and Cycle A2, and day 1 of Cycle B for a total of 3 doses during Course 2.
  Patients with an initially abnormal flow study, who show no evidence of obstructive hydrocephalus or compartmentalization on the repeat study, may begin intrathecal mafosfamide administration with the initiation of Regimen 1, Course 2. The frequency of intrathecal mafosfamide administration, for such patients, will be as outlined in Regimen 1, Course
  1.
Drug: Regimen 2, Course 1 — Cycle C1 (Days 1 - 21) Day 1: Prehydrate with D5W 1/2 NS + KCl 2 mEq/100 ml) at 2 times the hourly maintenance rate until the urine specific gravity is < 1.012.
  0 hrs: Mesna 6 mg/kg IV over 15 min. Dilute in 0.65 ml/kg IVF. 15 min: Vincristine 0.05 mg/kg IV push (Day 1 only)(max dose = 2 mg) 20 min: Cyclophosphamide 30 mg/kg IV over 30 min. 50 min: Post-chemotherapy hydration - D5 1/2 NS + KCl
  (1 mEq/100 ml) at twice the hourly maintenance rate for at least 24 hours. 3 hrs: Mesna 6 mg/kg IV in 0.65 ml/kg IVF over 15 min 6 hrs: Mesna 6 mg/kg IV in 0.65 ml/kg IVF over 15 min 9 hrs: Mesna 6 mg/kg IV in 0.65 ml/kg IVF over 15 min 12 hrs: Mesna 6 mg/kg IV in 0.65 ml/kg IVF over 15 min Day 2: Repeat day 1, but omit vincristine. Day 3: G-CSF 5 µg/kg/day subcutaneously, daily, until ANC is > 2000 on two consecutive days, post ANC nadir.
Drug: Regimen 2, Course, 1, Cycle C1 — Cycle C1, Weeks 2 and 3 Day 8: Vincristine 0.05 mg/kg IV push (max dose = 2 mg) Day 15: Vincristine 0.05 mg/kg IV push (max dose = 2 mg) Cycle C2 (Days 22-42) Drugs and doses are same as in Cycle C1. Cycle C2 begins following recovery from Cycle C1, but no sooner than day 21. Patients with delays in recovery beyond day 28 should have dose modificationsCycle D (Days 43 - 63) Etoposide 1.7 mg/kg, po qd x 21 days The dose will be diluted immediately prior to administration in juice or flavored syrup as per section 3.4.3. Each dose should be taken 1 hour before or 2 hours after a meal.
  Cycle D should begin following recovery from Cycle C2; however, it should begin no sooner than 21 days after the start of Cycle C2.
Drug: Regimen 2, Course 2 — Repeat Course 1 (Cycle C1, Cycle C2, and Cycle D) in patients with SD or better at the interim response evaluation. Chemotherapy should begin as soon as the patient has recovered from the toxicities of oral etoposide in cycle D, course 1. However, it should not begin any sooner than 7 days after the completion of Course 1.
Radiation: radiation therapy — Conformal Irradiation Patients who are initially M0 with a CR, PR, or SD to Regimen 1 induction chemotherapy (with or without second surgery) will receive local irradiation using conformal techniques. Treatment will commence within 2 weeks of completing Regimen 1 or second surgery. Treatment planning and technique may involve 3D conformal,IMRT, or proton planning and delivery, provided the guidelines regarding volume, dose,and normal tissue restrictions are honored.
  8.3.1 Fraction Size 180 cGy fractions will be used for all target volumes. 8.3.2 Fractionation Conventional fractionation will be used. Treatments will be given once daily, 5 days/week except for necessary interruptions secondary to medical or administrative reasons.

SUMMARY:
The purposes of this study are to find the highest dose of mafosfamide that can be given without causing severe side effects, to see how well the combination of these chemotherapy drugs and lower doses of radiation work to delay or stop the growth of the tumor, and to evaluate the pharmacokinetics (how the body handles) of Mafosfamide.

DETAILED DESCRIPTION:
All children in the study will receive Regimen 1 chemotherapy. Children whose tumor is limited to one area at the beginning of the study will go on to have radiation therapy and then Regimen 2 chemotherapy. Children whose tumor was found in more than one part of the brain or in the cerebrospinal fluid at the beginning of the study will discontinue their treatment on this protocol after Regimen 1 chemotherapy.

Regimen 1 Chemotherapy - Those children with a normal CSF flow study at the beginning of the study will receive Regimen 1 chemotherapy along with mafosfamide. Those children with an abnormal CSF flow study will receive Regimen 1 without mafosfamide and a repeat CSF flow study will be performed at the completion of the first 10 weeks of treatment. If the CSF study reflects normal CSF flow, then intrathecal mafosfamide will be given during the second 10 weeks of Regimen 1. Regimen 1 is divided into two courses. Each course lasts about 10 weeks, for a total of 20 weeks of treatment. During Regimen 1 the patient will receive three medications (cyclophosphamide, vincristine, and cisplatin) that are given through the central venous line. The patient will also receive one medication that is given by mouth (etoposide). Cyclophosphamide, vincristine, cisplatin, and etoposide are all anticancer drugs that have been useful in the treatment of brain tumors.

The experimental drug, mafosfamide, will be injected into the spinal fluid. This will be given through either a spinal tap, the Ommaya reservoir, or both. Alternating mafosfamide between the spinal tap and the Ommaya reservoir may improve how well the drug works by making sure it spreads throughout the spinal fluid. If the patient has a VP or VA shunt ( specialized devices that relieve the pressure inside the head that comes from a block in the normal flow of spinal fluid), then the patient will not receive an Ommaya reservoir, and all doses of mafosfamide will be given through a spinal tap only.

The starting dose of mafosfamide will be a dose that has been safely given to older children. If that dose does not cause severe side effects, the next group of patients will receive a higher dose of mafosfamide. If severe side effects occur, the next group of patients will receive a lower dose of mafosfamide

During and at the end of Regimen 1, the patient will be evaluated for response of the brain tumor to treatment. A second operation may be necessary to remove more of the brain tumor. Children whose tumor had spread at the time they began this study have completed treatment at this point. Children whose tumor had not spread at start of the study will begin radiation therapy, if their tumor appears to be unchanged or shrinking after Regimen 1.

Radiation Therapy - The dose, location, and timing of radiation will depend on the age of the child at diagnosis, the location of his/her tumor, and the response of his/her tumor to Regimen 1 chemotherapy. The radiation treatments used in this protocol are designed in an attempt to reduce some of the side effects that usually occur after standard radiation therapy.

The child will receive radiation using a new technology called "conformal radiation". Conformal radiation is designed to reduce the amount of normal brain tissue that is exposed to high doses of radiation.

Regimen 2 Chemotherapy - After radiation therapy,the patient will receive additional chemotherapy, which will last about 20 weeks. Regimen 2 chemotherapy is the same as the Regimen 1 chemotherapy, except that the patient will not be given the drugs cisplatin and mafosfamide.

Pharmacokinetic (PK) studies will be performed with a total of 2 doses of intrathecal mafosfamide. PK studies tell us how the patient's body handles the study drug, mafosfamide. Sampling times (times when we collect cerebrospinal fluid for the PK studies) will be prior to drug administration and at 10 minutes, 2 hours, and 4 hours following drug administration. These studies will be performed after one dose of drug given through the spinal tap and after one dose of drug is given through the Ommaya reservoir. The pharmacokinetic study is optional and you can choose not to allow these samples to be drawn. Refusing the pharmacokinetic study will not affect the patient's participation/treatment on this study.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

* Age: < 3 years.
* Histology: Patient must have a histologically confirmed primary intracranial CNS medulloblastoma/PNET or other embryonal tumor (medulloepithelioma, ependymoblastoma, neuroblastoma, pineoblastoma), atypical teratoid/rhabdoid tumor, intracranial germ cell tumor, or choroid plexus carcinoma. Patients with M+ ependymoma are also eligible.
* Performance Status: Karnofsky or Lansky >= 30%
* Bone Marrow Function: All patients must have a Hgb >= 10 g/dl, ANC >= 1,500/mm3, and a platelet >= 100,000/mm3. If the patient has a positive bone scan, then a pretreatment bone marrow aspirate and biopsy must be free of tumor.
* Hepatic/Renal Function: All patients must have adequate hepatic (total bilirubin < 1.5 mg/dl, SGPT < 5x normal), and renal (normal serum creatinine for age or technetium clearance > 40/ml/min/m2) function.
* Prior Therapy: Patients may not have received prior radiotherapy or chemotherapy, with the exception of steroids. Patients must not be receiving any other investigational agents. (Patients may receive investigational agents for supportive care 30 days after completion of all mafosfamide therapy.)
* Surgery: Patients must begin protocol therapy within 35 days of definitive surgery.
* Central Line: Patients must be willing to have a central line.
* CSF flow: Patients must be willing to have a CSF flow study to determine whether or not they will receive intrathecal chemotherapy. Patients without a VP or VA shunt must be willing to have an Ommaya reservoir if their CSF flow study does not show any evidence of obstruction to or compartmentalization of flow. Patients with obstruction to or compartmentalization of CSF flow on their initial flow study must be willing to have a repeat flow performed within the initial 10 weeks of induction therapy, ideally during weeks 8-10. If a repeat flow study shows resolution of obstruction or compartmentalization, patients are expected to begin intrathecal mafosfamide during Regimen 1 course 2 of therapy. Patients without a VP or VA shunt who have resolution of normal flow should additionally have an Ommaya reservoir placed.

Max Age: 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2000-04-04 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
To evaluate the feasibility, including expected disease progression, of delivering 20 weeks of systemic chemotherapy plus (IT) mafosfamide. | 20 weeks
  controlling the disease for at least 20 weeks.
To evaluate the safety and feasibility of a limited dose escalation schedule of IT mafosfamide in children < 3 years of age. | 5 years
  Toxicities observed during the last 18 weeks of IT therapy (prior to irradiation) together with the acute toxicities profiles observed during the initial 2 weeks of IT therapy will be used to derive the dose to be evaluated in the feasibility component of this study.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Blaney, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Brain Tumor Center at Duke University, Durham, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas

REFERENCES:
- [Derived] McLendon RE, Adekunle A, Rajaram V, Kocak M, Blaney SM. Embryonal central nervous system neoplasms arising in infants and young children: a pediatric brain tumor consortium study. Arch Pathol Lab Med. 2011 Aug;135(8):984-93. doi: 10.5858/2010-0515-OAR1. PMID 21809989